CLINICAL TRIAL: NCT00187369
Title: The Twin Birth Study: A Multicentre Randomised Controlled Trial Comparing Planned Vaginal Birth to Elective Caesarean Section of Twins More Than or Equal to 32 Weeks Gestation
Brief Title: The Twin Birth Study: A Trial Comparing Planned Vaginal Birth to Elective Caesarean Section of Twins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr Jon Barrett, Chief, Maternal-Fetal Medicine, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCT-63164; ISRCTN74420086
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2020-05-04 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Twin Pregnancy
Keywords: twins; twin births; multiples

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caesarean Section (Other): delivery by CS
  Interventions: Procedure: Method of Delivery
- Vaginal Birth (Other): delivery by VB
  Interventions: Procedure: Method of Delivery

INTERVENTIONS:
Procedure: Method of Delivery — CS or VB

SUMMARY:
For twin pregnancies at 32-38 weeks gestation, where twin A is head down, does a policy of planned caesarean section (CS) lower the likelihood of death or serious illness, during the first 28 days after birth, compared to a plan for vaginal birth (VB)?

DETAILED DESCRIPTION:
For twin pregnancies of 32-38 weeks gestation, where twin A is presenting cephalic, does a policy of planned CS decrease the likelihood of perinatal or neonatal mortality or serious neonatal morbidity, during the first 28 days after birth, compared to a policy of planned VB?

ELIGIBILITY:
Inclusion Criteria:

1. Women at 32 0/7 - 38 6/7 weeks gestation
2. Estimated fetal weight of each fetus 1500 - 4000 g
3. Both twins alive at time of randomization
4. Twin A is in cephalic position

Exclusion Criteria:

1. Monoamniotic twins
2. Lethal fetal anomaly of either fetus
3. Contraindication to labour or vaginal delivery for either twin
4. Previous participation in the Twin Birth Study

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2804 (Actual)
Dates: Start 2003-12; Primary Completion 2011-05 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon F Barrett, Principal Investigator — SHSC
Locations (1):
- Data Coordinating Centre/SHSC, Toronto, Ontario, Canada

REFERENCES:
- [Background] Barrett JF, Hannah ME, Hutton EK, Willan AR, Allen AC, Armson BA, Gafni A, Joseph KS, Mason D, Ohlsson A, Ross S, Sanchez JJ, Asztalos EV; Twin Birth Study Collaborative Group. A randomized trial of planned cesarean or vaginal delivery for twin pregnancy. N Engl J Med. 2013 Oct 3;369(14):1295-305. doi: 10.1056/NEJMoa1214939. PMID 24088091
- [Derived] Hochler H, Tevet A, Barg M, Suissa-Cohen Y, Lipschuetz M, Yagel S, Aviram A, Mei-Dan E, Melamed N, Barrett JFR, Fox NS, Walfisch A. Trial of labor of vertex-nonvertex twins following a previous cesarean delivery. Am J Obstet Gynecol MFM. 2022 Jul;4(4):100640. doi: 10.1016/j.ajogmf.2022.100640. Epub 2022 Apr 8. PMID 35398584
- [Derived] Dougan C, Gotha L, Melamed N, Aviram A, Asztalos EV, Anabusi S, Willan AR, Barrett J, Mei-Dan E. Cesarean delivery or induction of labor in pre-labor twin gestations: a secondary analysis of the twin birth study. BMC Pregnancy Childbirth. 2020 Nov 17;20(1):702. doi: 10.1186/s12884-020-03369-x. PMID 33203367
- [Derived] Aviram A, Lipworth H, Asztalos EV, Mei-Dan E, Melamed N, Cao X, Zaltz A, Hvidman L, Barrett JFR. Delivery of monochorionic twins: lessons learned from the Twin Birth Study. Am J Obstet Gynecol. 2020 Dec;223(6):916.e1-916.e9. doi: 10.1016/j.ajog.2020.06.048. Epub 2020 Jun 24. PMID 32592694
- [Derived] Aviram A, Lipworth H, Asztalos EV, Mei-Dan E, Cao X, Melamed N, Zaltz A, Anastasio HB, Berghella V, Barrett JFR. The worst of both worlds-combined deliveries in twin gestations: a subanalysis of the Twin Birth Study, a randomized, controlled, prospective study. Am J Obstet Gynecol. 2019 Oct;221(4):353.e1-353.e7. doi: 10.1016/j.ajog.2019.06.047. Epub 2019 Jun 27. PMID 31254526
- [Derived] Mei-Dan E, Asztalos EV, Willan AR, Barrett JF. The effect of induction method in twin pregnancies: a secondary analysis for the twin birth study. BMC Pregnancy Childbirth. 2017 Jan 6;17(1):9. doi: 10.1186/s12884-016-1201-8. PMID 28061767
- [Derived] Melamed N, Wong J, Asztalos E, Rosen H, Okby R, Barrett J. The Likelihood of Change in Fetal Presentation During the Third Trimester in Twin Pregnancies. Obstet Gynecol. 2015 Dec;126(6):1231-1236. doi: 10.1097/AOG.0000000000001128. PMID 26551181

RESULTS

PARTICIPANT FLOW:
Groups:
- Caesarean Section: delivery by caesarean section
  Method of Delivery: CS or VB
- Vaginal Birth: delivery by vaginal birth
  Method of Delivery: CS or VB
Period: Mothers
Arm/Group | Caesarean Section | Vaginal Birth
Started | 1398 | 1406
Included in the Study | 1393 | 1393
Completed | 1392 | 1392
Not Completed | 6 | 14
Period: Fetuses or Infants
Arm/Group | Caesarean Section | Vaginal Birth
Started | 2795 | 2812
Included in the Study | 2785 | 2786
Completed | 2783 | 2782
Not Completed | 12 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caesarean Section | Vaginal Birth | Total
Number analyzed (Participants) | 1393 | 1393 | 2786
Age, Customized [Count of Participants; unit: Participants]
  Maternal age >= 30 yr | 632 | 632 | 1264
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 1393 | 1393 | 2786
Parity >= 1 [Count of Participants; unit: Participants] | 857 | 856 | 1713
Previous cesarean section [Count of Participants; unit: Participants] | 100 | 97 | 197
Gestational age at randomization [Count of Participants; unit: Participants]
  <32 wk 0 days | 0 | 1 | 1
  32 wk 0 days to 33 wk 6 days | 475 | 477 | 952
  34 wk 0 days to 36 wk 6 days | 679 | 665 | 1344
  37 wk 0 days to 38 wk 6 days | 239 | 250 | 489
Chorionicity at birth [Count of Participants; unit: Participants] — Chorionicity was determined by means of ultrasonography
  Participants
    Dichorionic and diamnionic | 961 | 970 | 1931
    Monochorionic and diamnionic | 334 | 326 | 660
    Unknown | 98 | 97 | 195
Not in labor at randomization [Count of Participants; unit: Participants] — Population: Data was missing from one woman in the planned cesarean delivery
  Participants
    number analyzed (Participants) | 1392 | 1393 | 2785
    (all) | 1190 | 1159 | 2349
Membranes ruptured at randomization [Count of Participants; unit: Participants] | 83 | 76 | 159
National perinatal mortality in mother's country of residence [Count of Participants; unit: Participants] — Countries included in the study that had fewer than 15 deaths per 1000 births were Australia, Belgium, Canada, Chile, Croatia, Estonia, Germany, Greece, Hungary, Israel, the Netherlands, Oman, Poland, Qatar, Romania, Serbia, Spain, the United Kingdom, the United States, and Uruguay; those with 15 to 20 deaths per 1000 births were Argentina, Brazil, and Jamaica; and those with more than 20 deaths per 1000 births were Egypt and Jordan.
  Participants
    <15 deaths/1000 births | 724 | 730 | 1454
    15-20 deaths/1000 births | 596 | 591 | 1187
    >20 deaths/1000 births | 73 | 72 | 145

OUTCOME MEASURES:

1. Primary Outcome: Perinatal/Neonatal Mortality and/or Serious Neonatal Morbidity
Description: The primary outcome was a composite of fetal or neonatal mortality or serious neonatal morbidity.
Time Frame: until 28 days after delivery
Population: number of fetuses/infants
Measure: Count of Participants; unit: Participants
Groups:
- Planned Caesarean Section: delivery by CS or Method of Delivery: CS or VB
- Planned Vaginal Birth: delivery by VB or Method of Delivery: CS or VB
Arm/Group | Planned Caesarean Section | Planned Vaginal Birth
Number analyzed (Participants) | 2783 | 2782
Participants
  Composite primary outcome | 60 | 52
  Death | 24 | 17
  Fetal death | 13 | 9
  Neonatal death | 11 | 8
  Serious neonatal morbidity | 36 | 35

2. Secondary Outcome: Neonatal Morbidity
Description: Neonatal morbidity, excluding death of either twin
Time Frame: until 28 days after delivery
Measure: Count of Participants; unit: Participants
Groups:
- Planned Caesarean Section: delivery by caesarean section
  Method of Delivery: CS or VB
- Planned Vaginal Birth: delivery by vaginal birth
  Method of Delivery: CS or VB
Arm/Group | Planned Caesarean Section | Planned Vaginal Birth
Number analyzed (Participants) | 2759 | 2765
Participants
  Long bone fracture | 0 | 4
  Other bone fracture | 1 | 1
  Facial-nerve injury at 72 hr of age or discharge | 0 | 1
  Intracerebral hemmorrhage | 3 | 1
  Apgar score at 5 minutes less than 4 | 2 | 7
  Coma | 0 | 1
  Stupor or decreased response to pain | 2 | 0
  Hyperalert, drowsy, or lethargic | 9 | 7
  ≥2 seizures within 72 hr after birth | 3 | 3
  Assisted ventilation for ≥24 hr by means of endotr | 27 | 17
  Neonatal sepsis within 72 hours after birth | 1 | 2
  Meningitis within 72 hours after birth | 0 | 0
  Necrotizing enterocolitis | 1 | 3
  Broncho-pulmonary dysplasia (BPD) | 0 | 0
  Grade 3 or 4 intraventricular hemorrhage | 0 | 0
  Cystic periventricular leukomalacia | 2 | 0

3. Secondary Outcome: Death or Poor Neurodevelopmental Outcome of the Children at 2 Years of Age (Corrected for Gestational Age at Birth)
Description: Neurodevelopmental outcome will be assessed by the Ages and Stages Questionnaire (ASQ). The ASQ is a parent/parental caregiver-administered structured questionnaire that includes questions on 5 domains of development: communication, gross motor skills, fine motor skills, problem-solving skills, and personal-social skills. If the score for any 1 of the 5 domains is below the specific cutoff for the domain, the ASQ was considered abnormal.
Time Frame: 2 years
Population: Neurodevelopmental outcomes of children at 2 years of age (based on available two year data of the children).
Measure: Count of Participants; unit: Participants
Arm/Group | Planned Caesarean Section | Planned Vaginal Birth
Number analyzed (Participants) | 2320 | 2283
Participants
  Fetal or neonatal death | 24 | 17
  Death up to follow-up | 11 | 6
  Neurodevelopmental delay: number analyzed (Participants) | 2285 | 2260
  Neurodevelopmental delay | 104 | 110
  Cerebral palsy: number analyzed (Participants) | 2285 | 2260
  Cerebral palsy | 2 | 1
  Motor delay: number analyzed (Participants) | 2285 | 2260
  Motor delay | 62 | 78
  Cognitive delay: number analyzed (Participants) | 2320 | 2258
  Cognitive delay | 95 | 105

4. Secondary Outcome: Problematic Urinary or Faecal/Flatal Incontinence of Mothers at 2 Years Postpartum
Description: The occurrence of problematic urinary, faecal/flatal incontinence at 2 years following the birth will be determined by structured questionnaire
Time Frame: 2 years postpartum
Measure: Count of Participants; unit: Participants
Groups:
- Planned Caesarean Section: delivery by CS
  Method of Delivery: CS or VB
- Planned Vaginal Birth: delivery by VB
  Method of Delivery: CS or VB
Arm/Group | Planned Caesarean Section | Planned Vaginal Birth
Number analyzed (Participants) | 1155 | 1150
Participants
  Urinary incontinence | 187 | 250
  Problematic urinary incontinence | 93 | 140
  Fecal incontinence | 47 | 68
  Problematic faecal incontinence | 21 | 29
  Flatal incontinence | 180 | 224
  Problematic flatal incontinence | 68 | 82

5. Other Pre Specified Outcome: Baseline Characteristics - Gestational Age at Randomization
Time Frame: Basline
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Planned Caesarean Section | Planned Vaginal Birth
Number analyzed (Participants) | 1393 | 1393
weeks | 34.9 (1.8) | 34.9 (1.8)

6. Other Pre Specified Outcome: Baseline Characteristics - Estimated Fetal Weight
Time Frame: Basline
Population: Data were missing for the following characteristics: estimated fetal weight of the first twin (for two women in the planned-cesarean-delivery group and for two in the planned-vaginal-delivery group) and estimated fetal weight of the second twin (for two women in the planned-cesarean-delivery group and for one in the planned-vaginal-delivery group)
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Planned Caesarean Section | Planned Vaginal Birth
Number analyzed (Participants) | 1393 | 1393
grams
  First Twin: number analyzed (Participants) | 1391 | 1391
  First Twin | 2238 (424) | 2238 (419)
  Second Twin: number analyzed (Participants) | 1391 | 1392
  Second Twin | 2223 (413) | 2232 (422)

7. Other Pre Specified Outcome: Other Maternal Outcomes
Description: Maternal depression at 2 years postpartum; Breastfeeding at 2 years postpartum
Time Frame: 2 years postpartum
Population: Available data
Measure: Count of Participants; unit: Participants
Arm/Group | Planned Caesarean Section | Planned Vaginal Birth
Number analyzed (Participants) | 1155 | 1150
Participants
  Depression (EPDS >12) | 129 | 115
  Continuing breast feeding: number analyzed (Participants) | 1129 | 1124
  Continuing breast feeding | 110 | 144

8. Other Pre Specified Outcome: Other Maternal Outcomes
Description: Maternal quality of life at 2 years postpartum (scores were reported using a scale of 0-100 with '0' indicating maximum disability and '100' no disability);
Time Frame: 2 year postpartum
Population: Mean and standard deviation on available data. This is based on available maternal data at 2 years postpartum.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Planned Caesarean Section | Planned Vaginal Birth
Number analyzed (Participants) | 1141 | 1134
score on a scale
  Maternal quality of life (SF-36) Physical | 53.4 (7.0) | 53.2 (6.9)
  Maternal quality of life (SF-36) Mental | 47.9 (10.4) | 48.1 (10.8)

9. Other Pre Specified Outcome: Other Maternal Outcomes
Description: Maternal depression at 3 months; Problematic urinary or faecal/flatal incontinence at 3 months; Breastfeeding at 3 months
Time Frame: 3 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Planned Caesarean Section | Planned Vaginal Birth
Number analyzed (Participants) | 1285 | 1285
Participants
  >12 (probable depression) | 180 | 190
  ≥10 (possible depression | 298 | 306
  Experienced any urinary incontinence | 145 | 197
  Problematic urinary incontinence | 70 | 82
  Experienced faecal incontinence | 49 | 48
  Problematic faecal incontinence | 18 | 17
  Experienced incontinence of flatus | 205 | 145
  Problematic flatal incontinence | 62 | 79
  Breastfed either baby at any time | 1084 | 1110
  Stopped breastfeeding at <15 days | 32 | 45

10. Other Pre Specified Outcome: Other Maternal Outcomes
Description: Maternal quality of life at 3 months (scores were reported using a scale of 0-100 with '0' indicating maximum disability and '100' no disability); Maternal fatigue at 3 months (the scale combines 16 items to produce a Global Fatigue Index (GFI), which can range from 1 (no fatigue) to 50 (severe fatigue)); Maternal depression at 3 months was measured by the Edinburgh Postnatal Depression Scale, which measures how women have been feeling in the previous 7 days, with a score of >12 indicating depression (each answer is given a score of 0 to 3 based on the seriousness of the symptom. The total possible maximum depression score is 30). IIQ-7 at 3 months are validated questions about the impact of the incontinence (scores were reported using a scale of 0-100, with '0' indicating no impact at all and '100' greatly impacted).
Time Frame: 3 months postpartum
Population: Mean and standard deviation on available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Planned Caesarean Section | Planned Vaginal Birth
Number analyzed (Participants) | 1285 | 1285
units on a scale
  Maternal quality of life (SF-36) Physical: number analyzed (Participants) | 1258 | 1260
  Maternal quality of life (SF-36) Physical | 51.8 (7.1) | 51.6 (7.6)
  Maternal quality of life (SF-36) Mental: number analyzed (Participants) | 1258 | 1260
  Maternal quality of life (SF-36) Mental | 46.7 (10.9) | 46.0 (11.3)
  Global Fatigue Index score: number analyzed (Participants) | 1251 | 1251
  Global Fatigue Index score | 20.3 (8.8) | 20.8 (9.3)
  Edinburgh Postnatal Depression Scale: number analyzed (Participants) | 1283 | 1282
  Edinburgh Postnatal Depression Scale | 5.7 (5.6) | 5.9 (5.7)
  Incontinence Impact Questionnaire-7 (IIQ-7): number analyzed (Participants) | 70 | 82
  Incontinence Impact Questionnaire-7 (IIQ-7) | 20.48 (21.41) | 20.44 (20.50)

ADVERSE EVENTS:
Description: Fusion and adverse events were connected and baby. There were no serious adverse Maternal events.
Groups:
- Planned Caesarean Section-Mother; Planned Caesarean Section-Infants/Fetuses: delivery by CS or Method of Delivery: CS or VB
- Planned Vaginal Birth-Mother; Planned Vaginal Birth-Infants/Fetuses: delivery by VB or Method of Delivery: CS or VB
Arm/Group | Planned Caesarean Section-Mother | Planned Vaginal Birth-Mother | Planned Caesarean Section-Infants/Fetuses | Planned Vaginal Birth-Infants/Fetuses
All-Cause Mortality (participants affected / at risk) | 0/1392 | 0/1392 | 24/2783 | 17/2782
Serious Adverse Events (participants affected / at risk) | 0/1392 | 0/1392 | 0/2783 | 0/2782
Other Adverse Events (participants affected / at risk) | 0/1392 | 0/1392 | 0/2783 | 0/2782

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No